CLINICAL TRIAL: NCT05926622
Title: Clinical and Radiological Outcomes of Medacta Shoulder System
Brief Title: Clinical and Radiological Outcomes of Medacta Shoulder System FR
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P06.001.03
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Primary Osteoarthritis; Secondary Osteoarthritis; Rotator Cuff Tear Arthropathy; Rheumatoid Arthritis Shoulder; Avascular Necrosis; Fracture; Revision of Shoulder Arthroplasty
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Osteonecrosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a post-marketing surveillance on Medacta Shoulder System

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patient with one of the following diagnosis:

Primary osteoarthritis Secondary osteoarthritis Cuff tear arthropathy; insufficient rotator cuff Acute fracture (<21d) Rheumatoid or inflammatory arthritis Avascular necrosis Other posttraumatic condition Revision of shoulder arthroplasty

Exclusion Criteria:

* Patients with malignant diseases (at the time of surgery)
* Patients with proven or suspect infections (at the time of surgery)
* Patients with functional deficits other than dysfunction of the shoulder (at the time of surgery)
* Patients with known incompatibility or allergy to products materials (at the time of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring TSA and who are suitable to receive Medacta Shoulder System will be proposed to take part to the current post-marketing surveillance study during their pre-operative visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2037-03 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | 10 years
  Kaplan Meier method

SECONDARY OUTCOMES:
Clinical outcome evaluating Constant & Murley Score | 1, 2, 5 and 10 years
  Constant & Murley Score (CMS): The CMS is a multi-item functional scale assessing pain, ADL, ROM and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively
Functional outcome evaluating Oxford Shoulder Score | 1, 2, 5 and 10 years
  Oxford Shoulder Score (OSS): The Oxford Shoulder Score is a unidimensional score comprising 12 questions. Starting with 1 (best/fewest symptoms) to 5 (worst/most severe) which is awarded to correspond to the patient's symptoms. The total gives a minimum score of 12 and a maximum of 60. A higher score implies a greater degree of disability.
Radiographic performance of the implants evaluating presence of radiolucencies | 3 months, 1, 2, 5 and 10 years
  presence of radiolucencies
Patient evaluation quality of life | 1, 2, 5 and 10 years
  EQ-5D-5L: The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Typically it is calculated by assigning a numerical value to each response level (i.e., 1 for "no problems", 5 for "extreme problems"/"unable to") and summing these values across the five items, resulting in a score from 5 (no problems on any dimension) to 25 (extreme problems on all dimensions)
Adverse events | up to 10 years
  record of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Toussaint, Principal Investigator — Clinique Générale Annecy
Locations (1):
- Clinique Générale Annecy, Annecy, France

IPD SHARING:
Plan to Share IPD: No